CLINICAL TRIAL: NCT03585166
Title: Comparison of Efficacy and Nursing Between Laparoscopic Hepatectomy and Open Hepatectomy for Primary Liver Cancer
Brief Title: Nursing Fro Laparoscopic vs. Open Hepatectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zeng Li, Charge nurse, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: WHUH2018S002
Record Dates: First submitted 2018-04-24; First posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Liver Cancer; Liver Neoplasms
Keywords: Liver Cancer; laparoscopic hepatectomy; open hepatectomy
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic hepatectomy: laparoscopic hepatectomy for primary liver cancer
  Interventions: Procedure: lpaparoscopic hepatectomy
- open hepatectomy: open hepatectomy for primary liver cancer
  Interventions: Procedure: open hepatectomy

INTERVENTIONS:
Procedure: lpaparoscopic hepatectomy — laparoscopic hepatectomy： laparoscopic hepatectomy for hepatocellular carcinoma.
  Groups: laparoscopic hepatectomy
Procedure: open hepatectomy — open hepatectomy: open hepatectomy for hepatocellular carcinoma
  Groups: open hepatectomy

SUMMARY:
This study was divided into laparoscopic hepatectomy (observation group) and laparoscopic hepatectomy (control group).Compared two groups of age, sex, body mass index (BMI), tumor diameter, number of tumors (single/multiple), pathologic characteristics, HBsAg (positive/negative), liver function, AFP, Child - Pugh, grading, nursing method and comparison of two groups of patients after surgery (surgical incision length, intraoperative blood, intraoperative blood transfusion and transfusion volume, operation time) the number of cases of and postoperative rehabilitation (death cases, for the first time the meal time, anus exhaust time, analgesic bed, first time, the abdominal cavity drainage tube time, length of hospital stay, postoperative days and liver function index.Follow-up: the survival rates of the two groups were compared in six months, one year, two years, three years and five years.In this study, the initial selection of the minimum sample size of 30 cases, plus 20% inefficiencies, the final initial selection of 36 cases, and the later expansion of the sample size of 100 cases.The research date starts on October 1, 2017.

DETAILED DESCRIPTION:
Research design and methods:

This study was divided into laparoscopic hepatectomy (observation group) and laparoscopic hepatectomy (control group).Compared two groups of age, sex, body mass index (BMI), tumor diameter, number of tumors (single/multiple), pathologic characteristics, HBsAg (positive/negative), liver function, AFP, Child - Pugh, grading, nursing method and comparison of two groups of patients after surgery (surgical incision length, intraoperative blood, intraoperative blood transfusion and transfusion volume, operation time) the number of cases of and postoperative rehabilitation (death cases, for the first time the meal time, anus exhaust time, analgesic bed, first time, the abdominal cavity drainage tube time, length of hospital stay, postoperative days and liver function index.Follow-up: the survival rates of the two groups were compared in six months, one year, two years, three years and five years.In this study, the initial selection of the minimum sample size of 30 cases, plus 20% inefficiencies, the final initial selection of 36 cases, and the later expansion of the sample size of 100 cases.

Statistical methods: by means of SPSS 23.0 to analyze the data, all data after the normal test to choose the appropriate statistical methods, the normal distribution of measurement data in the two groups use surgery and postoperative recovery using two sets of samples t test, liver function index using analysis of variance, non-normal distribution using nonparametric test, count data chi-square test, P < 0.05 for the difference was statistically significant.Survival analysis was performed on two groups of patients.The research date starts on October 1, 2017.

ELIGIBILITY:
Inclusion criteria:

Hepatocellular carcinoma There was no distant metastasis in patients with malignant tumors. Exclusion criteria: primary tumor diameter > 10cm Thrombosis of portal or inferior vena cava carcinoma Severe organic disease or cirrhosis of the liver Laparoscopic transposition of the abdomen Concomitant coagulant function abnormal patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult, aged (18- N/A),male/femal,diagnosised with primary hepatoma, received surgical intervention(laparoscopic and open)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of complications of primary liver cancer treated by laparoscopic hepatectomy and laparoscopic hepatectomy,The questionnaire survey | Patients with hepatocellular carcinoma who were hospitalized together on October 1, 2017 were studied at the time point before discharge.
  The incidence of complications, in percent
The survival rate of primary liver cancer treated by laparoscopic hepatectomy and laparoscopic hepatectomy,Telephone pays a return visit | 1 month after discharge
  Survival rate, percent
The survival rate of primary liver cancer treated by laparoscopic hepatectomy and laparoscopic hepatectomy,Telephone pays a return visit | 3 month after discharge
  Survival rate, percent
The survival rate of primary liver cancer treated by laparoscopic hepatectomy and laparoscopic hepatectomy,Telephone pays a return visit | 6 month after discharge
  Survival rate, percent
The survival rate of primary liver cancer treated by laparoscopic hepatectomy and laparoscopic hepatectomy,Telephone pays a return visit | 1 year after discharge
  Survival rate, percent
The survival rate of primary liver cancer treated by laparoscopic hepatectomy and laparoscopic hepatectomy,Telephone pays a return visit | 2 year after discharge
  Death and recurrence
The survival rate of primary liver cancer treated by laparoscopic hepatectomy and laparoscopic hepatectomy,Telephone pays a return visit | 3 year after discharge
  Death and recurrence
The survival rate of primary liver cancer treated by laparoscopic hepatectomy and laparoscopic hepatectomy,Telephone pays a return visit | 5 year after discharge
  Survival rate, percent

SECONDARY OUTCOMES:
Comparison of oxygen uptake days between laparoscopic hepatectomy and laparoscopic hepatectomy for primary liver cancer, unit: day | Patients with liver cancer who are hospitalized on 1 October 2017 will be included in the study date.The study time is 1 year.
  Oxygen uptake days, per day
Comparison of ecg monitoring days between laparoscopic hepatectomy and laparoscopic hepatectomy for primary liver cancer Unit: day | Patients with liver cancer who are hospitalized on 1 October 2017 will be included in the study date.The study time is 1 year.
  Guardianship days, unit: days
Comparison of the number of replacement drainage bags for primary hepatocellular carcinoma between laparoscopic hepatectomy and laparoscopic hepatectomy, unit: number | Patients with liver cancer who are hospitalized on 1 October 2017 will be included in the study date.The study time is 1 year.
  Compare the number of times to replace the drainage bag, unit: number
Comparison of infusion days between laparoscopic hepatectomy and laparoscopic hepatectomy for primary liver cancer Unit: day | Patients with liver cancer who are hospitalized on 1 October 2017 will be included in the study date.The study time is 1 year.
  Infusion days, unit: days
Comparison of muscle injection times between laparoscopic hepatectomy and laparoscopic hepatectomy in primary liver cancer: times | Patients with liver cancer who are hospitalized on 1 October 2017 will be included in the study date.The study time is 1 year.
  Muscle injections,Unit: times
Comparison between laparoscopic hepatectomy and laparoscopic hepatectomy in primary hepatocellular carcinoma Unit: times | Patients with liver cancer who are hospitalized on 1 October 2017 will be included in the study date.The study time is 1 year.
  Number of subcutaneous injections Unit: times

CONTACTS AND LOCATIONS:
Overall Officials: Li Zeng, Principal Investigator — Department of Hepatobiliary,Union Hospital,Tongji Medical College, Huazhong University of Science and Technology, Wuhan 430022, China
Locations (1):
- Union hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No